CLINICAL TRIAL: NCT05796648
Title: Preparing a Food is Medicine Intervention to Promote Healthy Eating and Blood Pressure Control in Black Women with Hypertension and Obesity
Brief Title: Preparing a Food is Medicine Intervention to Promote Healthy Eating and Blood Pressure Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: University of Chicago (Other); Rush University (Other)
Responsible Party: Principal Investigator, Saria Lofton, Assistant Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0947; P50MD017349 (NIH)
Record Dates: First submitted 2022-12-13; First posted 2023-04-03 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-11

CONDITIONS: Hypertension; Obesity; Healthy Nutrition; Blood Pressure
MeSH Terms: conditions — Hypertension; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Food is Medicine approach (Experimental): Groups of 10 will attend a 12 week intervention that includes cooking classes, grocery delivery and nutrition education.
  Interventions: Behavioral: RN-CHeFRx

INTERVENTIONS:
Behavioral: RN-CHeFRx — The RN-CHeFRx trial to enhance dietary intake and blood pressure control in Black women with hypertension and obesity compared to usual care.

SUMMARY:
Hypertension and obesity are both major risk factors for cardiovascular disease (CVD), a leading cause of death for Black women in the United States. The investigators propose examining the feasibility and acceptability of the 12-week RN-CHeFRx (Real Nourishment and Cooking Healthy Food is Rx) intervention - grocery delivery, cooking classes, and nutrition education - for Black women with hypertension and obesity to improve nutritious eating habits and blood pressure control.

DETAILED DESCRIPTION:
The objective of this study is to conduct the RN-CHeFRx (Real Nourishment and Cooking Healthy Food is Rx) for 12 weeks among Black women who are obese and hypertensive living Chicago. We propose to 1) Pilot the RN-CHEFRx intervention and measures that will be used to assess blood pressure, BMI status, and sodium intake with 20 Black women diagnosed with hypertension and BMI ≥ 30. We will assess the efficacy of the evaluation tools to be used in a future clinical trial at three-time points (baseline, 12 weeks, and 6 months); and 2) Assess the feasibility and acceptability of the RN-CHeFRx intervention using interviews, surveys, and documentary analysis. Findings from this study will inform a larger efficacy trial of RN-CHeFRx to improve dietary behaviors and blood pressure control among Black women with hypertension and obesity.

ELIGIBILITY:
Inclusion Criteria:

* self-identified as Black or of African descent
* female
* ≥ 18 years old
* baseline blood pressure ≥130/85 or diagnosed with hypertension and BMI ≥ 30

Exclusion Criteria:

* inability to cook in their homes
* cognitive deficits impeding the ability to participate or provide informed consent
* current treatment for cancer
* liver or renal disease
* pregnancy
* lack of English language proficiency

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Number of participants who complete the 12 week intervention | Up to 12 weeks
  Completion will be measured by class attendance
Number of participants recruited | Up to 12 weeks
  Patients recruited, screened, eligible and consented to participate in the study
Number of participants who complete data collection visits | Baseline to 4 months
  Completion measured by participants completing surveys, blood pressure measurements, and those who provide blood biospecimens
Acceptability of the intervention | Up to 12 weeks
  Assessed via participant feedback
Change in mean blood pressures (mmHg) during intervention | Baseline to 12 weeks
  Change will be measured by comparing blood pressures from baseline to 12 weeks
dietary intake during intervention | Baseline to 12 weeks
  Dietary intake at baseline and 12 weeks

SECONDARY OUTCOMES:
Change in body weight during intervention | Up to 12 weeks
  Change will be measured by comparing body weight obtained at baseline and 12 weeks
Change in body weight at 6 months | 12 weeks to 24 weeks
  Change will be measured by comparing body weight (kg) obtained at 12 weeks and at 24 weeks.
Change in blood pressure at 6 months | 12 weeks to 24 weeks
  Change will be measured by comparing systolic and diastolic blood pressure at 12 weeks to 24 weeks
Dietary intake during post-intervention | 12 weeks to 24 weeks
  Dietary intake from 12 weeks to 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No